CLINICAL TRIAL: NCT05749198
Title: Non-invasive Assessment of Portal Hypertension Using Quantitative Magnetic Resonance Imaging
Brief Title: Portal Hypertension Using Magnetic Resonance Elastography
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Moon Young Kim, Professor, Yonsei University
Other Study IDs: CR317132
Record Dates: First submitted 2023-02-14; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Portal Hypertension; Magnetic Resonance Imaging
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRE — MRE was performed using a 3T system (Magnetom Skyra; Siemens, Erlangen, Germany) equipped with a combination of a 30-channel body and a 32-channel spine matrix coil.

SUMMARY:
This prospective study was conducted in a tertiary university hospital. The investigators researched the correlation between MRE-assessed stiffness of the liver and spleen and the Hepatic venous pressure gradient (HVPG) values. Furthermore, the investigator evaluated whether MRE-assessed stiffness reflected changes in portal hypertension (PH) after administering non-selective beta-blockers (NSBBs).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed liver cirrhosis
* requiring prophylactic treatment of esophageal varices

Exclusion Criteria:

* the coexistence of hepatocellular carcinoma
* refractory ascites who regularly underwent large-volume paracentesis
* the use of selective beta-blocker or carvedilol therapy for at least 4 weeks
* undergoing liver transplantation
* contraindication with magnetic resonance imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring prophylactic treatment of esophageal varices
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Change of liver stiffness and spleen stiffness by MRE | Change from baseline stiffness of MRE at 6 months
The change of portal pressure (HVPG) prior to and after treatment with NSBB | Change from baseline and at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No